CLINICAL TRIAL: NCT01042249
Title: The Effect of Pelvic Floor Muscle Training on Lower Urinary Tract Symptoms (LUTS) in Men With Stroke
Brief Title: Pelvic Floor Muscle Training(PFMT) on Lower Urinary Tract Symptoms (LUTS) in Men With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Fondation of 18.12.1981 (Other)
Responsible Party: Principal Investigator, Sigrid Tibaek, pt, Dr Med Sci, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-B-2009-069
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Male; Stroke; Urinary Incontinence
Keywords: PFMT; Stroke; LUTS; Men
MeSH Terms: conditions — Stroke; Urinary Incontinence; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Treated with Pelvic Floor Muscle Training in 12 weeks
  Interventions: Other: Pelvic Floor Muscle training
- Control (No Intervention): Receives standard rehabilitation after stroke

INTERVENTIONS:
Other: Pelvic Floor Muscle training — 12 week training program including home exercises
  Arms: Treatment

SUMMARY:
The aim of this study is to evaluate the effect of pelvic floor muscle training (PFMT) on Lower Urinary Tract Symptoms (LUTS) in men after stroke.

120 men with LUTS or increased LUTS after stroke is included and randomized into a treatment group or a control group. The subjects in the treatment group follows a 12 week standard PFMT program, while the control group is not given specific treatment of their LUTS but like the treatment group follows the standard rehabilitation program for stroke patient. Outcome are measured by

* 5 questionnaires
* Voiding diary
* 24-hour pad test
* pelvic floor muscle assessment test

ELIGIBILITY:
Inclusion Criteria:

1. Men, diagnosed with stroke clinical defined according World Health Organisation (WHO 1989) and confirmed by CT and MRI scan
2. Onset of last stroke ≥ 1 month
3. Normal cognitive function (minimal mental examination score > 25 ) (Folstein, Folstein et al. 1976).
4. LUTS according to ICS definition (Abrams, Cardozo et al. 2002), with start or aggravation in close relation to the stroke
5. Independent walking abilities indoor > 100 m with/without aids
6. Independence in toilet visits
7. Age > 18 years

Exclusion Criteria:

1. Prior history of LUTS surgery, pelvic surgery or trauma
2. More than 2 hospital diagnosed stroke
3. Other severe neurological diseases including dementia
4. Severe dysphasia
5. Severe psychiatric disease
6. Prostate cancer
7. Do not speak Danish or English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-02; Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
DAN-PSS-1 questionnaire | 2010-2012

SECONDARY OUTCOMES:
Pelvic Floor Muscle Assessment test | 2010-2012

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of physiotherapy and occupational therapy, Glostrup University Hospital, Copenhagen, Glostrup Municipality, Denmark